CLINICAL TRIAL: NCT04551872
Title: Personalizing Cardiovascular Health: A Population Approach to Promoting CVD Resistance and Resilience Among Individuals With Obesity
Brief Title: RESILIENCE: Personalizing Cardiovascular Health
Acronym: RESILIENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00104664
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Cardiovascular Risk Factor
Keywords: Obesity; Translating Duke Health; RESILIENCE; CVD; DUHS; Duke; Heart Disease
MeSH Terms: conditions — Obesity; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Obese High Risk (Experimental): 200 participants with BMI ≥30 and 10-year ASCVD risk ≥20%
  Interventions: Behavioral: Digital weight loss intervention
- Obese Low Risk (Experimental): 200 participants with BMI ≥30 and 10-year ASCVD risk <7.5%
  Interventions: Behavioral: Digital weight loss intervention
- Non-Obese High Risk (No Intervention): 100 participants with BMI 18-25 and 10-year ASCVD risk ≥20%
- Non-Obese Low Risk (No Intervention): 100 participants with BMI 18-25 and 10-year ASCVD risk <7.5%

INTERVENTIONS:
Behavioral: Digital weight loss intervention — Participants with obesity enter into a proven 6 month weight loss program that utilizes health coaching and goal-setting. It is a remote intervention that is delivered entirely over their phones. Participants will also receive a FitBit and electronic scale.
  Arms: Obese High Risk; Obese Low Risk

SUMMARY:
Obesity is a rapidly growing epidemic that is associated with the development of cardiovascular disease (CVD). However, some individuals with obesity appear to be resistant to CVD, and other individuals demonstrate resilience to obesity and CVD risk factors. The investigator's overall objective is to understand factors contributing to the heterogeneity of CVD resistance and resilience among individuals with obesity at Duke.

DETAILED DESCRIPTION:
The investigator aims to recruit participants with 4 phenotypes: 200 participants with obesity (BMI ≥ 30) and high 10-year ASCVD risk (≥20%), 200 participants with obesity (BMI ≥ 30) and low 10-year ASCVD risk (<7.5%), 100 participants with normal weight (BMI 18-25) and high 10-year ASCVD risk (≥20%), and 100 participants with normal weight (BMI 18-25) and low 10-year ASCVD risk (<7.5%). Clinical, behavioral, and molecular characteristics will be compared at baseline between the 4 groups to understand heterogeneity between obesity and risk for CVD, and participants with obesity will undergo a 6-month weight loss intervention. In individuals with obesity, clinical, behavioral, and molecular characteristics will be compared between baseline and 6 months to understand (a) predictors of response to the intervention and (b) how these factors change with weight loss. Differences in branched-chain amino acids will be compared between all groups, both at baseline and at 6 months (for those participants undergoing the digital-weight loss intervention). Other clinical, behavioral, metabolomic, genetic, and microbiome parameters will also be compared in an exploratory fashion. There may be possible risk of loss of confidentiality, but this risk is low and measures will be taken to minimize this risk.

Recruitment Sub-Study: We aim to determine optimal strategies to recruit participants into the study via electronic recruitment. We will identify potentially eligible participants within the Duke Electronic Health Record and reach out them via electronic means. Potentially eligible participants will be randomized in a 2x2 factorial fashion to receive personal email vs. MyChart message, and to different message content (1 of 4 types). We will analyze: a) which modality of introductory message delivery (MyChart vs personal email) will lead to greater engagement (as assessed by clicking on the study website page to get more information) b) which messages (altruism vs personal benefit vs scientific importance) will lead to greater engagement.

Consent Sub-Study: We aim to determine optimal strategies to consent participants into the study via e-consent portal. Potential participants who land on the study website will be randomized to consent via one of four methods, followed by a consent-comprehension quiz: a) video consent with study information provided by a representative patient, b) video consent with study information provided by the lead physician of the study, c) video consent with study information provided by animation/cartoon or d) text-based study information and consent (standard). We will analyze which type of consent form will lead to greater completion of consent forms and greater comprehension of the consent form.

Coronary Artery Calcium (CAC) Score Sub-Study: At baseline visit, a total of 300 participants (150 with obesity and 150 without obesity) will undergo CT testing to determine coronary artery calcium (CAC) score.

Basic Science Sub-Study: Thirty participants with obesity (15 high-risk for CV disease and 15 low-risk for CV disease) will participate in the basic science sub-study where additional blood will be drawn at baseline visit and at follow-up visit. This blood will be processed to isolate the endothelial colony forming cells and we will examine the effect of altered plasma branched chain amino acid (BCAA) levels on vascular function within these groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults 40-75 years old
* At least one clinic encounter at Duke with BMI record in the EHR within previous year
* Has a current primary care provider listed listed in EHR
* No prior history of ASCVD, as defined by ICD9, ICD10, and CPT codes for coronary artery disease, myocardial infarction, stroke, peripheral arterial disease, prior revascularization for coronary, cerebral, or peripheral arteries.
* Fall into 1 of 4 categories: 200 participants with obesity (BMI ≥ 30) and high 10-year ASCVD risk (≥20%), 200 participants with obesity (BMI ≥ 30) and low 10-year ASCVD risk (<7.5%), 100 participants with normal weight (BMI 18-25) and high 10-year ASCVD risk (≥20%), and 100 participants with normal weight (BMI 18-25) and low 10-year ASCVD risk (<7.5%).
* Have internet access
* Have an email address listed in the EHR
* Have access to MyChart
* Have a smartphone
* Be able to read and understand English

Exclusion Criteria:

* Participants "opted out" of being contacted for research in Maestro Care
* Pregnant at the time of enrollment or <12 months post-partum
* Prior bariatric surgery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Average branched-chain amino acid levels as measured by metabolomics analyses | Baseline
Change in branched-chain amino acid levels as measured by metabolomics analyses | Baseline, End of intervention (up to 6 months)

OTHER OUTCOMES:
Gut microbiome composition as measured by DNA sequencing | Baseline
Change in gut microbiome composition as measured by DNA sequencing | Baseline, End of intervention (up to 6 months)
Genetic markers as measured by whole exome sequencing of DNA from saliva | Baseline
Impact of branched-chain amino acids on tissue engineered blood vessel function as measured by monocyte adhesion | Baseline
Impact of branched-chain amino acids on tissue engineered blood vessel function as measured by foam cell formation | Baseline
Change in impact of branched-chain amino acids on tissue engineered blood vessel function as measured by monocyte adhesion | Baseline, End of intervention (up to 6 months)
Change in impact of branched-chain amino acids on tissue engineered blood vessel function as measured by foam cell formation | Baseline, End of intervention (up to 6 months)
Average levels of inflammation measured by hs-CRP | Baseline
Change in average levels of inflammation measured by by hs-CRP | Baseline, End of intervention (up to 6 months)
Average lipid profile as measured by total cholesterol | Baseline
Change in lipid profile as measured by total cholesterol | Baseline, End of intervention (up to 6 months)
Average lipid profile as measured by HDL | Baseline
Change in lipid profile as measured by HDL | Baseline, End of intervention (up to 6 months)
Average lipid profile as measured by LDL | Baseline
Change in lipid profile as measured by LDL | Baseline, End of intervention (up to 6 months)
Average blood glucose control as measured by HbA1c | Baseline
Change in blood glucose control as measured by HbA1c | Baseline, End of intervention (up to 6 months)
Average blood glucose control as measured by fasting glucose | Baseline
Change in blood glucose control as measured by fasting glucose | Baseline, End of intervention (up to 6 months)
Average blood glucose control as measured by blood insulin level | Baseline
Change in blood glucose control as measured by blood insulin level | Baseline, End of intervention (up to 6 months)
Average coronary artery calcium score as measured by CT testing | Baseline
Change in coronary artery calcium score as measured by CT testing | Baseline, End of intervention (up to 6 months)
Engagement as measured by percent of invitees viewing study-information page | End of study, up to 2 years
Best consent strategy as measured by percent of invitees signing the consent form | End of study, up to 2 years
Best consent strategy as measured by average score on Informed Consent Form comprehension quiz | End of study, up to 2 years
  7 multiple choice questions, best outcome is 7/7 (100%), worst outcome is 0/7 (0%)

CONTACTS AND LOCATIONS:
Overall Officials: Neha Pagidipati, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No